CLINICAL TRIAL: NCT03168035
Title: A Phase 1 Dose-Escalation and Pharmacokinetic Study of NC-4016 in Patients With Advanced Solid Tumors or Lymphoma
Brief Title: Study of NC-4016 in Patients With Advanced Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NanoCarrier Co., Ltd. (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NC-4016-001; NCT01999491 (obsolete NCT alias)
Record Dates: First submitted 2017-04-03; First posted 2017-05-30 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Advanced Cancer; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — NC-4016

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NC-4016 (Experimental): Dose Escalation Group: NC-4016 will be administered as 2-hour intravenous infusion once every 3 weeks. Initial dose level 15 mg/m2. The dose level of NC-4016 in subsequent cohorts determined by the toxicity profile of the previous cohort, and dose level increased to 25, 30, 40, 60, and 80 mg/m2 or higher at each subsequent cycle until the highest dose level is reached or DLT prohibits further dose-level escalation. Dose level 1 will be the starting dose level (DL). If 2 out of the first 3 patients enrolled at DL1 experience a DLT during Cycle 1 or Cycle 2,then the next cohort of patients will be enrolled at DL0 (10 mg/m2).
  Dose Expansion Group: Maximum tolerated dose from Dose Escalation Group
  Interventions: Drug: NC-4016

INTERVENTIONS:
Drug: NC-4016 — Dose Escalation Group Starting Dose: 15 mg/m2 by vein on Day 1 of a 21 Day cycle.
  Dose Expansion Group Starting Dose: Maximum tolerated dose from Dose Escalation Group.

SUMMARY:
The goal of this clinical research study is to find the highest tolerated dose of NC-4016 that can be given to patients with advanced solid tumors or lymphoma. The safety of the drug will also be studied.

DETAILED DESCRIPTION:
Study Groups:

If participants are found to be eligible to take part in this study, they will be enrolled in either a dose escalation group or the dose expansion group.

Dose Escalation:

If participants are in a dose escalation group, they will be assigned to a dose level based on when they joined this study. Up to 6 dose levels of NC-4016 will be tested and at least 3 patients will be enrolled at each dose level. The first group of participants will receive the lowest dose level of NC-4016. Each new group will receive a higher dose of NC-4016 than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of NC-4016 is found.

Dose Expansion:

If participants are in the dose expansion group, they will receive NC-4016 at the highest dose that was tolerated in the escalation groups.

Study Drug Administration:

Each study cycle is 21 days.

On Day 1 of each cycle, you will receive NC-4016 by vein over 2 hours.

Participants will be given standard drugs to help decrease the risk of side effects. They may ask the study staff for information about how the drugs are given and their risks.

If participants have a severe side effect, their dose of study drug may be delayed.

Study Visits:

On Day 1 of each cycle:

* Participants will have a physical exam.
* Their vital signs (blood pressure, heart rate, breathing rate, and temperature) will be monitored every 20 minutes during the infusion and 1 hour after the end of the infusion during Cycle 1 and right before and at the end of the infusion for all other cycles.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* Participants will have a neurological exam and electromyogram.
* Participants will have an EKG before the start of the infusion, at the end of the infusion, and 1 hour after the end of the infusion (Cycle 1 and 2 only). After Cycle 1, Participants will only have 1 EKG before dosing.

On Days 8 and 15 of each cycle, blood (about 3 teaspoons) will be drawn for routine tests.

On Day 2 of Cycle 1 participants will have an EKG corresponding to the 24 hour PK testing.

Every 3 cycles (every 9 weeks):

* Participants will have an x-ray, CT, MRI, or PET scan to check the status of the disease.
* If participants have lymphoma, they will have a bone marrow biopsy to check the status of the disease.
* Participants will have a nerve conduction evaluation.
* If the doctor thinks it is needed, blood (about 1 teaspoon) will be drawn for tumor marker testing.

PK Testing:

Blood (about 1 teaspoon each time) will be drawn for pharmacokinetic (PK) testing. PK testing measures the amount of study drug in the body at different time points.

* On Day 1 of Cycles 1 and 3, blood will be drawn before, then at 0.5, 1, and 2 hours during the infusion, and then 9 more times up to 12 hours after participants receive the study drug (13 draws total each day).
* On Days 2, 3, 4, 6, 8, and 15 of Cycles 1 and 3, blood will be drawn 1 time after participants receive the study drug.
* On Day 1 of Cycles 2 and Cycle 4, blood will be drawn 1 time before participants receive the study drug.

Urine Collection:

Urine will be collected for PK testing at the following time points during Cycles 1 and 3:

* Before participants receive the study drug
* 0-2 hours (during the infusion)
* 2-4 hours after they received the study drug
* 4-8 hours after they received the study drug
* 8-12 hours after they received the study drug
* 12-24 hours after they received the study drug

Participants will collect their urine at home over 24 hours during the following times after they received the study drug:

* Days 1-2
* Days 2-3
* Days 7-8
* Days 14-15
* Days 21-22

The study doctor will provide participants with urine collection bottles. Urine samples will contain a very small amount of platinum from the study drug. This is not considered to be a risk, but as a precaution, the urine collection containers should only be handled by participants, and the containers will be labeled as a "Bio-Hazard".

If participants have a severe side effect, they may have extra tests until the side effects have gotten better.

Length of Study:

Participants may continue taking the study drug for as long as they are benefitting. Participants will be taken off study early if the disease gets worse, intolerable side effects occur, they develop new health problems, their doctor thinks that it is no longer in their best interest to receive the study drug, or if they are unable to follow study directions.

Participants' participation on the study will be over after the end-of-dosing visit.

End-of-Dosing Visit:

Within 28 days after the last dose of NC-4016 participants will:

* Have a physical exam.
* Have a neurological exam and an electromyogram.
* Have a chest x-ray.
* Have an x-ray, CT scan, MRI scan, or PET scan, or a bone marrow biopsy if they have lymphoma, to check the status of the disease.
* Blood (about 3 teaspoons) and urine will be collected for routine tests.
* Have an EKG and an ECHO or MUGA.
* If the doctor thinks it is needed, blood (about 1 teaspoon) will be drawn for tumor marker testing.

This is an investigational study. NC-4016 is not commercially available or FDA approved. It is currently being used for research purposes only. The study doctor can explain how NC-4016 is designed to work.

Up to 40 participants will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Have signed written informed consent prior to the initiation of any study-specific procedures
2. Be a male or female 18 years or older
3. Have a histologically or cytologically confirmed diagnosis of advanced solid tumor or lymphoma, or primitive hepatocarcinoma with radiological diagnosis
4. Have advanced or metastatic disease refractory to standard curative or palliative therapy or contraindication to standard therapy
5. Have an ECOG performance status of 0-2
6. Have adequate bone marrow reserve: a. Absolute neutrophil count at least 1.5 x 10^9/L, b. Platelet count at least 100 x 10^9/L, and c. Hemoglobin at least 10 g/L (transfusion is allowed to achieve hemoglobin of 10 g/L)
7. Have adequate liver function: a. Total serum bilirubin no more than 1.5 x upper limit of normal (ULN), and b. Alanine aminotransferase and aspartate aminotransferase<= 2.5 x ULN or <= 5.0 x ULN in case of documented hepatic metastasis
8. Have adequate renal function: glomerular filtration rate >=50 mL/min (calculated according to the formula of Cockcroft and Gault)
9. Be reasonably recovered from preceding major surgery as judged by the investigator or no major surgery within 4 weeks prior to the start of Day 1 treatment
10. Have a negative pregnancy test for females at screening, preferably done within 1 week before Day 1 of treatment (not applicable to patients with bilateral oophorectomy and/or hysterectomy)
11. Be willing to abstain from heterosexual activity or practice physical barrier contraception from study entry to 6 months after the last day of treatment

Exclusion Criteria:

1. Have peripheral neuropathy of Grade 3 or Grade 4 at screening, according to National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE)v4.03, 14 June 2010 scale; or TNSc score greater than 4
2. Have an interval from previous neurotoxic platinums of less than 6 months and/or from previous other neurotoxic drugs less than 3 months (eg, taxanes) unless reasonably recovered from all grades of neurotoxicity as judged by the investigator
3. Have a history of thrombocytopenia with complications including hemorrhage or bleeding >= Grade 2 using NCI CTCAE v4.03, 14 June 2010 that required medical intervention or any hemolytic condition or coagulation disorders that would make participation unsafe in the opinion of the investigator
4. Have unresolved toxicity from previous treatment or previous investigational agents; excluding alopecia. Clinical judgment by the investigator is allowed to determine if grade 1 fatigue at screening is residual toxicity from prior treatment or is a symptom of the patient's general condition or disease. The investigator and medical monitor will discuss the eligibility of patients with baseline toxicity
5. Have known hypersensitivity to Pt compounds
6. Have received investigational agents or systemic anticancer agents (other than neurotoxic compounds) within 14 days of Day 1 of treatment, or 28 days for those agents with unknown elimination half-lives, or known elimination half-lives greater than 50 hours; or 6 weeks for mitomycin C or for nitrosourea agents
7. Is pregnant or breast-feeding
8. Have signs or symptoms of end organ failure, major chronic illnesses other than cancer, or any severe concomitant conditions which, in the opinion of the investigator, make it undesirable for the patient to participate in the study, or which could jeopardize compliance with the protocol
9. Have experienced any of the following within the 6-month period prior to screening: angina pectoris, coronary artery disease or cerebrovascular accident, transient ischemic attack, cardiac failure with known ejection fraction less than 40%, or cardiac arrhythmia requiring medical therapy
10. Have known hepatitis B or C, or human immunodeficiency virus infection
11. Is unwilling or unable to comply with study procedures, or is planning to take a vacation for 7 or more consecutive days during the treatment phase of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of NC-4016 | 21 days
  MTD defined as the highest dose level at which no more than 1 of 6 dose limiting toxicity (DLT) evaluable patients experience a DLT during Cycle 1 of dosing. DLT determined by NCI CTCAE v4.03, 14 June 2010.

SECONDARY OUTCOMES:
Cmax | During the First 4 Cycles of Treatment (each cycle is 21 days)
  calculated for all patients using noncompartmental analysis
Tmax | During the First 4 Cycles of Treatment (each cycle is 21 days)
  calculated for all patients using noncompartmental analysis
AUC | During the First 4 Cycles of Treatment (each cycle is 21 days)
  calculated for all patients using noncompartmental analysis
T1/2 | During the First 4 Cycles of Treatment (each cycle is 21 days)
  calculated for all patients using noncompartmental analysis
CL | During the First 4 Cycles of Treatment (each cycle is 21 days)
  calculated for all patients using noncompartmental analysis
Vss | During the First 4 Cycles of Treatment (each cycle is 21 days)
  calculated for all patients using noncompartmental analysis
Vz | During the First 4 Cycles of Treatment (each cycle is 21 days)
  calculated for all patients using noncompartmental analysis
Excretion Profile of Total and Free (Ultrafiltrate) Platinum (Pt) | Cycle 1 and Cycle 3 (each cycle is 21 days)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org